CLINICAL TRIAL: NCT07211048
Title: Early Exploratory Clinical Study of CD19-targeted Gene Injection (LCAR02) in Patients With Relapsed/Refractory B-cell Lymphoma
Brief Title: Anti CD19 Gene Therapy for B-cell Lymphoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2025ky481
Record Dates: First submitted 2025-09-30; First posted 2025-10-07 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-09

CONDITIONS: B-cell Lymphoma
Keywords: B-cell lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti CD19 Gene Therapy for B-cell Lymphoma (Experimental)
  Interventions: Drug: Anti-CD19 gene injection

INTERVENTIONS:
Drug: Anti-CD19 gene injection — Intravenous infusion of Anti-CD19 gene injection （three dosage groups）

SUMMARY:
This is an open label, single-site, dose-escalation study in up to 18 participants with treatment of relapsed/refractory B-cell lymphoma. This study aims to evaluate the safety and efficacy of the treatment with an Anti- CD19 gene injection

ELIGIBILITY:
Inclusion Criteria:

* (1)Age 18 years or older, any gender; (2)Patients diagnosed with any of the following conditions: diffuse large B-cell lymphoma (DLBCL), germinal center or activated B-cell type; primary cutaneous DLBCL; primary mediastinal (thymic) large B-cell lymphoma; ALK-positive anaplastic large B-cell lymphoma; high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements; high-grade B-cell lymphoma; T-cell-rich B-cell lymphoma; transformed follicular lymphoma; or any aggressive B-cell lymphoma arising from indolent lymphoma; follicular lymphoma; mantle cell lymphoma; large cell transformation of CLL. Patients must have previously received at least second-line standard treatment and either did not achieve remission or relapsed after remission; (3) For B-cell lymphoma patients, according to the preliminary assessment, staging, and response evaluation recommendations for Hodgkin and non-Hodgkin lymphomas (2014 edition), there must be at least one measurable lesion at baseline, which is defined as a lymph node lesion with a long diameter >15 mm or an extranodal lesion with a long diameter >10 mm, diagnosed by PET-CT or CT imaging; (4) B-cell lymphoma patients must have tumor cells confirmed CD19 positive by immunohistochemistry; (5) Adequate vital organ function: liver function meeting: ALT ≤3×ULN, AST ≤3×ULN; serum creatinine ≤140 μmol/L; total bilirubin ≤2×ULN, or ≤3×ULN in patients with Gilbert's syndrome; hemodynamically stable as determined by echocardiography or multi-gated radionuclide angiography (MUGA) with left ventricular ejection fraction (LVEF) ≥45%; no active pulmonary infection, and percutaneous arterial oxygen saturation ≥92% without supplemental oxygen; (6) ECOG performance status: 0-2; (7) Expected survival of more than 3 months; (8) Female and male participants of childbearing potential must agree to use reliable and effective contraception from the time of signing the informed consent form until 2 years after receiving LCAR02 infusion (excluding natural family planning methods).

Exclusion Criteria:

* (1) Patients who have experienced central nervous system diseases or pathological changes within 6 months before screening, including but not limited to: stroke, cerebrovascular accident, aneurysm, epilepsy, convulsions, aphasia, severe traumatic brain injury, dementia, Parkinson's disease, cerebellar diseases, organic brain syndrome, or mental disorders.

  (2) Patients with malignant tumors other than B-cell lymphoma. (3) Patients who received vaccines or B-cell targeted therapy within 4 weeks before screening.

  (4) Patients with systemic autoimmune diseases or immunodeficiency. (5) Patients with grade 2-4 acute graft-versus-host disease (GVHD) or moderate to severe chronic GVHD within 4 weeks before screening.

  (6) Patients with relatively severe heart disease, such as angina, myocardial infarction, heart failure, or arrhythmia.

  (7) Patients with a history of severe allergies to the drugs or excipients used in the clinical study or investigational drugs.

  (8) Patients with active hepatitis B, HCV antibody positivity, HIV antibody positivity, or positive for syphilis.

  (9) Patients with active infections requiring intravenous antibiotics or hospitalization.

  (10) Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-03-20 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | up to 1 years
  Total number, incidence and severity of adverse events (AEs) in patients of LCAR1901 infusion. The AEs will be assessed according to the 2019 Consensus on Cytokine Release Syndrome and Immune-cell-associated Neurotoxicity published by the American Society of Transplantation and Cell Therapy (ASTCT), the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 and EBMT 2019 consensus.
The persistence, accumulation, and migration of anti-CD19 gene injection | up to 1 years
  Assessing the trafficking of anti-CD19 gene injection in the peripheral blood at the time of each infusion as well as at each time of follow-up by Quantitative Real-time Polymerase Chain Reaction or flow cytometry. Peripheral blood will be collected prior to the initial infusion and will be set as baseline.

SECONDARY OUTCOMES:
Complete response (CR) rate | up to 1 year
  Evaluation of disease efficacy according to the 2014 Lugano criteria. CR rate is defined as the proportion of patients who have achieved CR assessed by investigators.
Objective response rate (ORR) | up to 1 year
  ORR is defined as the proportion of patients who have achieved CR and partial response (PR) assessed by investigators.
Duration of Response (DOR) | up to 1 year
  DOR is defined as the date of their first CR or PR (which is subsequently confirmed) to PD assessed by investigators, or death regardless of cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Provincial Hospital, Hefei, Anhui, China